CLINICAL TRIAL: NCT01084668
Title: A Post-marketing Observational Study of the Quality of Life in Adalimumab Treated Psoriasis Patients Failing Other Biologic DMARDs Over a Period of 1 Year (QUALITY)
Brief Title: Quality of Life in Adalimumab Treated Psoriasis Patients Failing Other Biologic Disease Modifying Anti-rheumatic Drugs
Acronym: QUALITY
Status: Completed | Type: Observational
Sponsor: Abbott (Industry)
Collaborators: Assign Data Management and Biostatistics GmbH (Other)
Responsible Party: Sponsor
Other Study IDs: P10-708
Record Dates: First submitted 2010-02-28; First posted 2010-03-10 (Estimated); Results first posted 2012-05-30 (Estimated); Last update posted 2012-06-29 (Estimated); Status verified 2012-06

CONDITIONS: Psoriasis Chronic
Keywords: moderate to severe chronic plaque psoriasis; adalimumab; Psoriasis Area and Severity Index (PASI); Disease Life Quality Index (DLQI); Nail Psoriasis Severity Index (NAPSI); biologic disease modifying anti-rheumatic drug (BDMARD); antibodies; monoclonals

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Adalimumab: Participants with moderate to severe chronic plaque psoriasis treated with adalimumab after biologic disease modifying anti-rheumatic drug (BDMARD) failure

SUMMARY:
The aim of this post-marketing observational study (PMOS) was to obtain further data on long-term safety, efficacy, and quality of life outcomes for adalimumab in routine clinical use in participants with moderate to severe chronic plaque psoriasis after unsustainable clinical response to other biologic disease modifying anti-rheumatic drugs (BDMARDs). There are few data so far showing the effects of switching from other BDMARDs to adalimumab in patients with moderate to severe chronic plaque psoriasis. This study was designed to evaluate the long-term effectiveness of adalimumab in participants with moderate to severe chronic plaque psoriasis using the Psoriasis Area and Severity Index (PASI) in participants previously treated with efalizumab, infliximab, or etanercept and who either never achieved satisfactory response, achieved satisfactory response initially but lost it over time, or discontinued treatment due to intolerance/side effect(s) or other reasons, for example after regular stop of etanercept.

DETAILED DESCRIPTION:
This was a non-interventional PMOS conducted in a prospective, single-country, multicenter format to assess the quality of life of psoriasis patients taking adalimumab as prescribed by their physician in accordance with the terms of the local marketing authorization with regard to dose, population, and indication. The prescription of adalimumab was clearly separated from the decision to include the participant in this study. No procedures other than standard of care were to have been performed. Visits were non-interventional and timing of participant appointments was left to each physician. After therapy initiation, visits occurred over 12 months usually close to Weeks 4, 12, 24, 36, and 52 for a total of 6 visits (Visits 1 through 6 including Screening). Because participant visits were left to the physician, participant failure to meet the suggested visit weeks did not constitute a breach of the protocol.

ELIGIBILITY:
Inclusion Criteria:

* Patients for whom adalimumab therapy is indicated and has been prescribed according to the product label
* Patients aged 18 years and older
* Unsatisfactory response to prior BDMARDS (efalizumab, infliximab, etanercept) in patients with moderate to severe chronic plaque psoriasis or achievement of satisfactory response initially, but loss over time or discontinuation of treatment due to intolerance/side effects(s) or other reasons e.g. restart after regular stop of etanercept
* Patients must fulfill Austrian Treatment Recommendations for use of BDMARD in psoriasis (chest X-ray and purified protein derivative [PPD] skin test negative for tuberculosis)
* Patient is willing to consent to data being collected and provided to Abbott
* Patient must be able and willing to self-administer Pen injections or have a qualified person available to administer Pen injections

Exclusion Criteria:

* Patients who meet contraindications as outlined in the latest version of the Humira-Pen Summary of Product Characteristics (SPC)
* Patients who do not meet the criteria for the use of BDMARDs of the Austrian Treatment Recommendations
* Patients participating in another study or clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hospital, Dermatology
Sampling Method: Non-Probability Sample
Enrollment: 46 (Actual)
Dates: Start 2008-11; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Astrid Dworan-Timler, MD, Study Director — Abbott Austria
Locations (9):
- Austria (9):
  - Site Reference ID/Investigator# 27435, Feldkirch
  - Site Reference ID/Investigator# 27436, Graz
  - Site Reference ID/Investigator# 38445, Graz
  - Site Reference ID/Investigator# 27443, Linz
  - Site Reference ID/Investigator# 27442, Vienna
  - Site Reference ID/Investigator# 27440, Vienna
  - Site Reference ID/Investigator# 27437, Vienna
  - Site Reference ID/Investigator# 27439, Vienna
  - Site Reference ID/Investigator# 23309, Wels

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 46 participants were screened for this PMOS at 9 study sites in Austria. One participant did not meet entry criteria (screening failure), and 45 participants were enrolled and received treatment with adalimumab in the study.
Pre-assignment Details: Three participants were excluded from the database because they had been treated with adalimumab prior to their Visit 1. Statistical analysis has been performed for the 42 participants included in the All Treated population.
Period: Overall Study
Arm/Group | Adalimumab
Started | 42 (Three participants who took Humira prior to study entry have been excluded from the database.)
Completed | 33
Not Completed | 9
Not completed — Lack of Efficacy | 5
Not completed — Withdrawal by Subject | 2
Not completed — Pregnancy | 1
Not completed — Non-compliance | 1

BASELINE CHARACTERISTICS:
Arm/Group | Adalimumab
Number analyzed (Participants) | 42
Age Continuous [Mean (Standard Deviation); unit: years] | 47.1 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 27
Region of Enrollment [Number; unit: participants]
  Austria | 42

OUTCOME MEASURES:

1. Primary Outcome: Psoriasis Area and Severity Index (PASI) Score
Description: Psoriasis Area and Severity Index (PASI) score is based on assessment of erythema (reddening), induration (plaque thickness), desquamation (scaling), and area affected as observed on the day of examination. The score ranges from 0 (best outcome) to 72 (worst outcome).
Time Frame: Inclusion visit (Week 0), Week 4, Week 36, Week 52
Population: Analysis was performed on the All Treated population using an observed case approach. PASI score was assessed at Weeks 0, 4, 36, and 52 in 41, 36, 28, and 27 participants, respectively.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- All Treated: Participants with moderate to severe chronic plaque psoriasis treated with adalimumab after biologic disease modifying anti-rheumatic drug (BDMARD) failure
Arm/Group | All Treated
Number analyzed (Participants) | 42
units on a scale
  Week 0 | 15.5 (11.4)
  Week 4 | 7.6 (4.5)
  Week 36 | 2.5 (5.2)
  Week 52 | 2.0 (4.9)

2. Primary Outcome: Reduction in Psoriasis Area and Severity Index Score of at Least 75% (PASI75)
Description: PASI75 is the number of participants who achieved at least a 75% reduction (improvement) from baseline in PASI score at Week 52 (final visit). PASI score is based on assessment of erythema (reddening), induration (plaque thickness), desquamation (scaling), and area affected as observed on the day of examination. The score ranges from 0 (best outcome) to 72 (worst outcome).
Time Frame: Inclusion visit (Week 0) to Week 52
Population: Analysis was performed on the All Treated population using an observed case approach. PASI response was assessed in 26 participants at Week 52.
Measure: Number; unit: participants
Arm/Group | All Treated
Number analyzed (Participants) | 26
participants | 23 (4.9)

3. Secondary Outcome: Dermatology Life Quality Index (DLQI) Score
Description: Dermatology Life Quality Index (DLQI) Score is a participant-reported outcome consisting of a set of 10 questions regarding the degree to which the participant's skin has affected certain behaviors and quality of life over the last week. Responses to each are: very much, a lot, a little, or not at all. The DLQI score ranges from 0 (best) to 30 (worst).
Time Frame: Inclusion visit (Week 0), Week 4, Week 36, Week 52
Population: Analysis was performed on the All Treated population using an observed case approach. DLQI score was assessed at Weeks 0, 4, 36, and 52 in 36, 34, 26, and 27 participants, respectively.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- All Treated: Participants with moderate to severe chronic plaque psoriasis treated with adalimumab after biologic disease modifying anti-rheumatoid drug (BDMARD) failure
Arm/Group | All Treated
Number analyzed (Participants) | 42
units on a scale
  Week 0 | 13.8 (8.3)
  Week 4 | 7.2 (5.6)
  Week 36 | 2.2 (3.4)
  Week 52 | 2.2 (4.8)

4. Secondary Outcome: Nail Psoriasis Severity Index (NAPSI) Score
Description: The nails are graded for nail matrix psoriasis and nail bed psoriasis. The sum of these two scores is the total score for that nail. Per nail, the NAPSI score ranges from 0 (no nail psoriasis) to 4 (most severe nail psoriasis).
Time Frame: Inclusion visit (Week 0), Week 4, Week 36, and Week 52
Population: Analysis was performed using an observed case approach. For the All Treated population, NAPSI was assessed at Weeks 0, 4, 36, and 52 in 34, 30, 24, and 25 participants, respectively. For the Subgroup with nail psoriasis, NAPSI was assessed at Weeks 0, 4, 36, and 52 in 18, 16, 12, and 13 participants, respectively.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Subgroup With Nail Psoriasis: Subgroup of participants with nail psoriasis and a NAPSI score greater than 0 for at least 1 study visit
Arm/Group | All Treated | Subgroup With Nail Psoriasis
Number analyzed (Participants) | 42 | 18
units on a scale
  Week 0 | 15.4 (24.0) | 29.0 (26.5)
  Week 4 | 14.9 (22.9) | 28.0 (25.0)
  Week 36 | 4.0 (9.6) | 7.9 (12.6)
  Week 52 | 4.0 (7.8) | 7.7 (9.5)

5. Secondary Outcome: Tolerability and Safety Assessed by Collection and Classification of Adverse Reactions
Description: Tolerability and safety were assessed by collecting adverse events during the course of the study up to 70 days following the last dose of physician-prescribed adalimumab. The number of participants experiencing a serious or non-serious adverse event is summarized. See the Reported Adverse Event section for details.
Time Frame: From the time of participant consent until 70 days after last dose of study drug
Population: Analysis was performed on the All Treated population.
Measure: Number; unit: participants
Arm/Group | All Treated
Number analyzed (Participants) | 42
participants
  Non-serious adverse events | 8
  Serious adverse events | 1

ADVERSE EVENTS:
Time Frame: Up to 1 year (from the time of participant consent through the final Week 52 visit) plus 70 days following administration of the last dose of physician-prescribed study treatment.
Arm/Group | Adalimumab
Serious Adverse Events (participants affected / at risk) | 1/42
Other Adverse Events (participants affected / at risk) | 8/42
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Adalimumab (N=42)
Ligament rupture (Injury, poisoning and procedural complications) | 1 (2)
Arthroscopic surgery (Surgical and medical procedures) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Adalimumab (N=42)
Acute tonsillitis (Infections and infestations) | 2
Nasopharyngitis (Infections and infestations) | 2
Injection site pain (General disorders) | 1
Injection site reaction (General disorders) | 1
Injection site urticaria (General disorders) | 1
Tooth fracture (Injury, poisoning and procedural complications) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1
Psoriasis (Skin and subcutaneous tissue disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Hypertension (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Abbott requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. Abbott requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if Abbott needs to secure patent or proprietary protection.